CLINICAL TRIAL: NCT04344132
Title: Pre- vs. Postoperative Scalp Block for Pain Control After Supratentorial Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Federico Bilotta, Principal investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: URom
Record Dates: First submitted 2020-03-30; First posted 2020-04-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Supratentorial Neoplasms
MeSH Terms: conditions — Supratentorial Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Scalp Block — standard practice of controll the pain after surgery. Block of the nerve emergences.

SUMMARY:
Study was designed to evaluate optimal timing for selective scalp block in patients undergoing general anesthesia for supratentorial craniotomy.Pain score assessed by visual analog scale (VAS) preoperatively (baseline) and after extubation at 2, 6, 12 and 24 hours; time first request of a patient for rescue analgesia; intraoperative anesthetics and opioids consumption; awakening time; perioperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years),
* presenting with supratentorial brain tumors scheduled for elective craniotomy under general anesthesia

Exclusion Criteria:

* history of allergic reactions on local anesthetics;
* ASA status ≥ 3;
* depressed consciousness in pre- or postoperative period;
* aphasia (as investigators were not able to obtain VAS score).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-20 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale score at 24 h after surgery | up to 24 hours
  Visual Analogue Scale ranging from 0 (no pain) to 10 (worst imaginable pain),

SECONDARY OUTCOMES:
Visual Analogue Scale score at 0 | Baseline
  Visual Analogue Scale ranging from 0 (no pain) to 10 (worst imaginable pain)
Visual Analogue Scale score at 2 hours | up to 2 hours
  Visual Analogue Scale ranging from 0 (no pain) to 10 (worst imaginable pain)
Visual Analogue Scale score at 6 hours | up to 6 hours
  Visual Analogue Scale ranging from 0 (no pain) to 10 (worst imaginable pain)
Visual Analogue Scale score at 12 hours | up to 12 hours
  Visual Analogue Scale ranging from 0 (no pain) to 10 (worst imaginable pain)
time first request of a patient for rescue analgesia | during surgery
intraoperative anesthetics | during surgery time
  (and opioids consumption)
awakening time | time from the end of surgery to awekening
changes in hemodynamics at mayfiled headfraom positioning | surgery
  changes in term of blood pressure
changes in hemodynamics at mayfiled headfraom positioning | surgery
  changes in heart rate

REFERENCES:
- [Background] Bebawy JF, Bilotta F, Koht A. A modified technique for auriculotemporal nerve blockade when performing selective scalp nerve block for craniotomy. J Neurosurg Anesthesiol. 2014 Jul;26(3):271-2. doi: 10.1097/ANA.0000000000000032. No abstract available. PMID 24492515
- [Background] Tsaousi GG, Logan SW, Bilotta F. Postoperative Pain Control Following Craniotomy: A Systematic Review of Recent Clinical Literature. Pain Pract. 2017 Sep;17(7):968-981. doi: 10.1111/papr.12548. Epub 2017 Feb 23. PMID 27996204